CLINICAL TRIAL: NCT03693274
Title: Mindfulness to Improve Functional Outcomes in Patients With Fibromyalgia or Central Sensitization: A Pilot Feasibility Study
Brief Title: Mindfulness to Improve Functional Outcomes in Patients With Fibromyalgia or Central Sensitization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator leaving institution.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jenna Walters, Assistant Professor of Anesthesiology and Pain Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 180985
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Chronic Pain; Fibromyalgia; Central Sensitisation
MeSH Terms: conditions — Chronic Pain; Fibromyalgia | interventions — Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Course (Experimental): Patient will be provided usual care for chronic pain at the Interventional Pain Clinic at Vanderbilt University Medical Center and will also be given access to BreatheAware for Pain Management, a 16- week web-based mindfulness course.
  Interventions: Behavioral: BreathAware for Pain Management
- Usual Care (No Intervention): Patient will be provided usual care for chronic pain at the Interventional Pain Clinic at Vanderbilt University Medical Center.

INTERVENTIONS:
Behavioral: BreathAware for Pain Management — Patients will be given access to a BreathAware, a 16- week web-based mindfulness course, which will be initiated at their enrollment. BreathAware is a self-paced course comprised of 2-3 minute lessons delivered via video, audio and technology-based guided instruction, and is available on a phone or tablet.
  Arms: Mindfulness Course

SUMMARY:
The primary aim of the study will be to determine the feasibility of utilizing a web-based mindfulness program in adult patients with chronic pain with a diagnosis of fibromyalgia or central sensitization.

DETAILED DESCRIPTION:
Chronic pain has a substantial economic cost and rate of impairment. Patients who suffer from fibromyalgia and other pain conditions leading to central sensitization have limited treatment options. The only medications currently approved by the Food and Drug Administration (FDA) for the treatment of fibromyalgia includes pregabalin, milnacipran and duloxetine. The International Association for the Study of Pain (IASP) also recommends the implementation of an exercise program and cognitive behavioral therapy. A previous meta-analysis found weak evidence to support Mindfulness-Based Stress Reductions (MBSR) in fibromyalgia patients, however more robust clinical studies are needed. In the midst of an opioid crisis, MBSR provides a safer alternative for the treatment of chronic pain. Unfortunately, an instructor lead MBSR program is both costly and largely unavailable in rural areas of the country. This web-based mindfulness program provides a treatment option for patients who would otherwise, not have access to alternative medicine therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30-65
* Patients with a diagnosis of fibromyalgia or central sensitization for greater than 6 months who are referred to the Interventional Pain Clinic

Exclusion Criteria:

* Patients on greater than 120 morphine equivalents per day
* Patients with untreated psychological illness
* Patients already enrolled in ongoing trials involving pain management and treatment interventions
* Patients currently undergoing treatment at the Osher Center for Integrative Health or patients with previous or current training in mindfulness.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Feasibility: Number of participants who complete the study | 17 weeks
  Number of participants who complete the study

SECONDARY OUTCOMES:
Change in mean Five Facet Mindfulness Questionnaire (FFMQ) score | Baseline and 17 weeks
  Comparison of mean score of FFMQ at baseline and 17 weeks of study participation. FFMQ is a self administered 39 item validated comprehensive instrument for assessing different aspects of mindfulness. Respondents rate statements according to how true the statement is to them on a scale of 1 (never or very rarely true) to 5 (very often or always true). Total scores are between 39 and 195 and higher scores indicate greater mindfulness.
Change in median Patient Reported Outcomes Measurement Information Systems-29 (PROMIS_29) score | Baseline and 17 weeks
  Comparison of mean PROMIS-29 score at baseline and 17 weeks of study participation.
  The PROMIS-29 (version 2) is a self administered validated instrument to assess seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. In addition, pain intensity is measured with a single item on an 11-point numeric scale (NPRS) that ranges from 0 to 10. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean more of the specific scale's construct, which may indicate a desirable or an undesirable outcome.
Change in Pain Catastrophizing Scale (PCS) | Baseline and 17 weeks
  Comparison of mean PCS score at baseline and 17 weeks of study participation. The PCS is measured with a self-administered questionnaire. The Pain Catastrophizing Scale is a 13-item inventory that measures 3 elements of the perception of the intensity of pain (rumination, magnification, feeling helpless). Participants indicate the degree to which they agree with statements related their pain by selecting 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree, 4 = all the time. There are three subscale scores assessing rumination, magnification and helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel.
Global Change | 17 weeks
  Global change measured by Patient Global Impression of Change (PGIC). The PGIC evaluates aspects of patients health and assesses if there has been an improvement or decline. The patient reports change in activity limitations, symptoms, emotions, and overall quality of life on scale from 1 (No change) to 7 (a great deal better), and the degree of change on a scale from 0 (much better) to 10 (much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Walters, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No